CLINICAL TRIAL: NCT01568411
Title: A Phase 1, Fixed-Sequence, Two-Period, Open-Label Drug-Drug Interaction Study to Assess the Effect of an Inhibitor of Cytochrome P450 Isoenzyme 3A4 and Permeability Glycoprotein 1 on the Pharmacokinetics of TD-1211
Brief Title: A Fixed-Sequence, Two-Period, Open-Label Drug-Drug Interaction Study to Assess the Effect of an Inhibitor of Cytochrome P450 Isoenzyme 3A4 and Permeability Glycoprotein 1 on the Pharmacokinetics of TD-1211
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0089
Record Dates: First submitted 2012-03-23; First posted 2012-04-02 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Healthy
Keywords: None - normal volunteers
MeSH Terms: interventions — 3-(8-(2-(cyclohexylmethyl(2,3-dihydroxypropionyl)amino)ethyl)-8-azabicyclo(3.2.1)oct-3-yl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TD-1211 (Active Comparator)
  Interventions: Drug: TD-1211
- TD-1211+ itraconazole (Active Comparator)
  Interventions: Drug: TD-1211+ itraconazole

INTERVENTIONS:
Drug: TD-1211 — Period 1
  Arms: TD-1211
Drug: TD-1211+ itraconazole — Period 2
  Arms: TD-1211+ itraconazole

SUMMARY:
This study will examine the effect of an inhibitor of cytochrome P450 isoenzyme 3A4 (CYP3A4) and permeability glycoprotein 1 (P gp) (200 mg itraconazole) on the PK disposition of a 10 mg tablet of TD- 1211 administered orally to fasted subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written, signed informed consent
2. Male and female subjects 18 to 50 years of age (inclusive)
3. Body mass index 19 to 30 kg/m2 (inclusive), and weigh at least 55 kg
4. No clinically important abnormal physical findings at the screening or Period 1, Day -1 examinations
5. Normal blood pressure (BP) and heart rate (HR). These will be measured after resting seated or supine for approximately 5 minutes. Normal BP is defined as 90 to 140 mm Hg systolic and 50 to 85 mm Hg diastolic. Normal HR is defined as 45 to 90 beats per minute
6. Negative for hepatitis B virus (HBV), hepatitis C virus (HCV), and human immunodeficiency virus (HIV) antibody within the last 3 months (documentation must be provided for confirmation)
7. No clinically relevant abnormalities in the results of Screening or Period 1, Day -1 laboratory evaluations
8. Ability to communicate effectively with the Investigator and to comply with all study requirements, restrictions, and direction of the clinic staff
9. For women of childbearing potential, documentation of a negative serum pregnancy test at Screening and a negative urine pregnancy test on Period 1, Day -1. Female subjects should not be breast feeding. All female subjects of childbearing potential must be using a highly effective method of birth control during the study and for at least 1 month after completion of study drug dosing. A highly effective method of birth control is defined as one that results in a low failure rate (i.e., <1% per year) when used consistently and correctly, such as condom + diaphragm, condom + spermicide, diaphragm + spermicide, or IUD with documented failure rate of <1% per year, or oral/injectable/implanted hormonal contraceptives used in combination with an additional double barrier method, or sexual abstinence. Women are considered to be not of childbearing potential if they have had a total hysterectomy or bilateral tubal ligation or are at least 2 years postmenopausal
10. All male subjects must agree to use a highly effective method of birth control with partners of childbearing potential during the study and for 1 month after study dosing

Exclusion Criteria:

1. Have evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, endocrine, pulmonary, GI, cardiovascular, hepatic, psychiatric, or neurological disease
2. Any condition possibly affecting drug absorption (e.g., previous surgery on the GI tract [including removal of parts of the stomach, bowel, liver, gall bladder, or pancreas])
3. Any other condition that, in the opinion of the Investigator, would confound or interfere with study participation; evaluation of safety, tolerability, or PK of the investigational drug; or prevent compliance with the study protocol
4. Have participated in another clinical trial of an investigational drug (or medical device) within 30 days (or 5 half lives of the investigational drug if longer than 30 days) prior to Screening, or are currently participating in another trial of an investigational drug (or medical device), or intending to participate in another trial of an investigational drug (or medical device) before completion of all scheduled safety evaluations in this trial
5. Unwilling to abstain from ingestion of caffeine or xanthine containing products (e.g., tea, coffee, chocolate, cola, etc.) beginning 48 hours before the dosing of study medication (Day 1) until the final PK sample in each period
6. History of hypersensitivity to drugs with a clinically significant reaction
7. Any history of alcoholism or drug abuse (in the past year) or positive screen for drugs of abuse or alcohol at Screening or Day -1 of each period.
8. Unwilling to abstain from alcohol beginning 48 hours prior to study dose administration (Day 1) until the collection of the final PK sample in each period.
9. Use or have used tobacco containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, etc.) within 6 months prior to Screening
10. Consumed grapefruit and/or grapefruit containing juice within 14 days, or apple or orange juice within 7 days prior to admission to the unit on Period 1, Day -1
11. Unwilling to abstain from ingestion of grapefruit, orange or apple juice throughout the duration of the study including the washout period.
12. Unwilling to abstain from any strenuous physical exercise (such as weight training, aerobics) 48 hours before the screening examination and 72 hours prior to study drug administration (Day 1) until collection of the final PK sample in each period
13. Acute illness (GI illness, infection [e.g., influenza] or known inflammatory process) on screening and/or admission to the clinical research unit for Period 1
14. Use of prescription drugs or any chronic over the counter medication including herbals within 7 days (or 14 days if the drug is a potential inducer or inhibitor of CYP3A4 or P gp [e.g., St John's Wort, rifampin, cyclosporine, or ritonavir]) or five half lives (whichever is longer) prior to Period 1, Day -1 or required continuing use during study participation, with the following exceptions:

    * Routine vitamins or minerals
    * Contraceptives and hormone replacement therapy (HRT)
    * A daily dose of acetaminophen (up to 1000 mg) or ibuprofen (up to 400 mg) if required on study
15. Have donated blood or blood components within the 8 weeks prior to Screening. The investigator should instruct subjects who participate in this study not to donate blood or blood components for 8 weeks after the completion of the study
16. Have an abnormal screening ECG indicating a second or third degree AV block, or one or more of the following: QRS >110 msec, QTc F >450 msec, PR interval >240 msec. Any rhythm other than sinus rhythm, which is interpreted by the investigator to be clinically significant
17. Personal or family history of congenital long QT syndrome or family history of sudden death
18. Known hypersensitivity towards or intolerance of TD 1211, itraconazole, or their formulation excipients contained in TD 1211 or itraconazole
19. Previous participation in another trial of TD 1211
20. Subjects who, for any reason, are deemed by the investigator to be inappropriate for this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Differences in pk parameters | 96 hours
  Assess the effect of CYP3A4 and P gp inhibition with itraconazole on the PK disposition of a single oral dose of TD-1211
  Endpoints included plasma PK parameters for TD-1211:
  * AUC
  * Cmax
  * Tmax
  * t1/2
  * CL/F
  * Vz/F

SECONDARY OUTCOMES:
Number of subjects with adverse events | 96 hours
  Assess the safety and tolerability of a single dose of TD-1211 when administered with an inhibitor of CYP3A4 and P gp

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Icon Development Services, San Antonio, Texas, United States